CLINICAL TRIAL: NCT06637995
Title: Product Surveillance Registry (PSR) - Nerve Integrity Monitoring (NIM) Vital Cohort
Brief Title: Product Surveillance Registry; Ear, Nose &Amp; Throat - NIM Vital Cohort
Acronym: PSR-ENT
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: PSR ENT - NIM Vital Cohort
Record Dates: First submitted 2024-09-23; First posted 2024-10-15 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Intracranial Surgery; Extracranial Surgery; Intratemporal Surgery; Extratemporal Surgery; Neck Surgery; Spine Surgery; Thoracic Surgery; Upper Extremity Surgery; Lower Extremity Surgery
Keywords: Nerve Monitoring; EMG Monitoring; Nerve Integrity
MeSH Terms: interventions — Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Device: Intraoperative Nerve Monitoring — Observational data collection from Locating, Stimulating, and Monitoring target nerves during a surgical procedure (clinician standard of care)

SUMMARY:
The purpose of this study is to confirm clinical safety and performance of Medtronic's NIM Vital™ System and accessories when used as intended in a real-world setting.

DETAILED DESCRIPTION:
Ongoing clinical investigation for the purpose(s) of:

* Providing continuing evaluation and periodic reporting of safety and effectiveness of Medtronic market-released products for their intended use
* Obtaining real-world performance and safety information from a global network of hospitals, clinics, and clinicians intended to represent the range of clinical environments in which Medtronic products are used
* Supporting post-market surveillance activities and post-approval studies that are initiated by Medtronic, regulated by local governments, or are conducted to fulfill government and/ or regulatory authority requests
* Obtaining clinical evidence to guide the development and improvement of medical devices, therapies, device guidelines, and patient services/solutions
* Providing clinical data to support health economics and clinical outcomes research

Enrollment for this study is ambispective, and subjects can be enrolled up to 60 days before or after the baseline procedure. There is no scheduled follow-up visit, however, if a reportable event occurs, patients will be followed until resolution or up to 6 months following the procedure. Total duration for study participants is anticipated to be 1 visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative (LAR) provides authorization and/or consent per institution and geographical requirements.
* Patient has or is intended to receive or be treated with an eligible Medtronic product
* Patient is consented within the enrollment window of the therapy received, as applicable

Exclusion Criteria:

* Patient who is, or is expected to be, inaccessible for follow-up
* Participation is excluded by local law
* Patient is currently enrolled or plans to enroll in concurrent drug/device study that may confound the PSR results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical procedures using the NIM Vital™ system and accessories for locating and monitoring, including stimulation, of cranial, spinal, peripheral motor and mixed motor-sensory nerves and registering electromyography (EMG) responses during surgery.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Adverse Event Rate | From enrollment to resolution of AE, or up to 6months following baseline procedure.
  Rate of adverse events caused directly by the NIM Vital™ System and/or accessories by determination and quantification of safety related complications.

SECONDARY OUTCOMES:
Device Performance | During baseline procedure
  Incidence of successful location, monitoring, and stimulation of target nerve, open airway for patient ventilation and EMG monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitatsklinikum Halle (Saale), Halle, Germany

IPD SHARING:
Plan to Share IPD: No